CLINICAL TRIAL: NCT05980520
Title: Taurine Supplementation Improves Core Symptoms in Children With Autism Spectrum Disorders: an Exploratory Randomized, Double-blinded, Controlled Trial
Brief Title: Study on the Treatment of Taurine in Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guizhou Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20230702
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
Keywords: autism spectrum disorders; children; taurine
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taurine treatment group (Experimental): Taurine combined with behavioral rehabilitation therapy
  Interventions: Dietary Supplement: Taurine+corn starch+white sugar; Behavioral: Behavioral rehabilitation therapy
- Placebo group (Placebo Comparator): Placebo combined with behavioral rehabilitation therapy
  Interventions: Dietary Supplement: Corn starch+white sugar; Behavioral: Behavioral rehabilitation therapy

INTERVENTIONS:
Dietary Supplement: Taurine+corn starch+white sugar — Taurine granules mixed with corn starch and white sugar, 0.4g in 1 bag, taken orally. One time dosage: 1 bag each time for 1-2 years old, 3 times a day, 1.5 bags each time for 3-5 years old, 3 times a day, 2 bags each time for 6-8 years old, 3 times a day, 2.5-3 bags each time for 9-13 years old, 3 to 4 bags each time for children and adults over 14 years old, 3 times a day. The use of taurine is strictly in accordance with the specifications of Chinese Pharmacopoeia.
  Arms: Taurine treatment group
Dietary Supplement: Corn starch+white sugar — 0.4g in 1 bag, taken orally. One time dosage: 1 bag each time for 1-2 years old, 3 times a day, 1.5 bags each time for 3-5 years old, 3 times a day, 2 bags each time for 6-8 years old, 3 times a day, 2.5-3 bags each time for 9-13 years old, 3 to 4 bags each time for children and adults over 14 years old, 3 times a day.
  Arms: Placebo group
Behavioral: Behavioral rehabilitation therapy — Structured training courses which included: visual arrangement, routine, environmental arrangement, program schedule, personal work system consists of five parts. The course is designed and implemented by qualified behavioral rehabilitators who have worked for more than 5 years, with the participation of parents. The daily training time is about 6-8 hours, and the total intervention time is not less than 40 hours per week.

SUMMARY:
In the treatment of autism spectrum disorders (ASD), medication is only an adjunct, and the main treatment modalities are education and behavioral therapy. People with autism incur huge medical and educational costs, which puts a great financial burden on families.Taurine is one of the abundant amino acids in tissues and organs, and plays a variety of physiological and pharmacological functions in nervous, cardiovascular, renal, endocrine and immune systems. A large number of studies have shown that taurine can improve cognitive function impairment under various physiological or pathological conditions through a variety of mechanisms, taurine can increase the abundance of beneficial bacteria in the intestine, inhibit the growth of harmful bacteria, and have a positive effect on intestinal homeostasis. This study intends to analyze the effect of taurine supplementation on ASD, and explore the possible mechanism by detecting intestinal symptoms, intestinal flora, markers of oxidative stress and clinical symptoms of ASD.

DETAILED DESCRIPTION:
Autism spectrum disorders (ASD) are the most common disabling disorders in childhood and are characterized by social difficulties, stereotyped behavior, narrow interests and paresthesia. In recent years, the prevalence of ASD has been increasing year by year, and the latest epidemiology in the United States shows that the prevalence of ASD is 1/44. The previous multi-center epidemiological survey of ASD in children in China showed that the prevalence of ASD in children aged 6-12 in China was about 0.7%, and the lifetime medical and non-medical expenses of ASD patients ranged from $1.4 million to $2.4 million. The survey showed that the disease burden of ASD in children aged 0-6 in Guizhou Province was between 60,000 and 80,000 yuan/year/person. ASD has become a major public health problem affecting children's health due to its high prevalence rate, disability rate and heavy disease burden, which has brought huge economic and social burden to families and society of children with ASD. At present, ASD has been listed as the leading disabling disease among mental diseases, bringing serious burden to families and society, and ASD has become a major public health problem affecting children's health.

At present, there are no specific drugs to improve the core symptoms of ASD, and education and behavioral therapy are mainly focused on early intervention to obtain the best results. Although effective behavioral interventions can significantly improve the core symptoms of children with ASD, a significant proportion of children with ASD still have residual functional disabilities. Therefore, the research and development of new treatment methods for children with ASD has become a hot and difficult problem. Children with ASD are prone to multiple nutrients due to poor eating habits, gastrointestinal symptoms and food allergies, and the addition of key nutrients is expected to become one of the important adjuvant treatments for children with ASD. The project team established a national children's ASD multi-center research cohort and built a children's ASD biobank under the financial support of the National Health Commission. A case-control (117:119) study using 1H-NMR metabolomics to detect urine samples of children with ASD showed lower taurine levels in the ASD group compared to the healthy control group. In recent years, taurine deficiency has been linked to neurological disorders or symptoms such as neurodegenerative diseases, stroke, epilepsy, and diabetic neuropathy. In addition, animal and clinical experiments have found that taurine supplementation has certain therapeutic effects on neurological diseases including Angelman behavior sign, fragile X behavior sign, sleep-wake disorder, stroke, attention deficit hyperactivity disorder, tic disorder, and taurine supplementation can improve anxiety symptoms and cognitive ability of mice. In previous animal intervention experiment, taurine supplementation on the basis of VPA autism model in rats during pregnancy was found to improve ASD-like behavior in offspring. However, there is a lack of population-based evidence in children with ASD.

Taurine is widely distributed in brain, spinal cord, heart, muscle cells and retina, and is one of the more abundant amino acids in almost all tissues and organs. A large number of studies have shown that taurine can protect a variety of tissues and organs from oxidative stress damage. Taurine can also ameliorate cognitive impairment in a variety of physiological and pathological conditions through a variety of mechanisms, including reducing neuroinflammation, up-regulating Nrf2 expression and antioxidant capacity, activating Akt/CREB/PGC1α signaling pathway to further enhance mitochondrial biosynthesis, synaptic function, and reducing oxidative stress. A large number of studies have shown that compared with healthy controls, the blood levels of oxidative stress markers in children with ASD are reduced or increased to varying degrees, and are thought to be related to the formation of stereotypical behaviors of ASD. Whether taurine can improve the core symptoms of ASD by reducing oxidative stress damage remains unclear, and human studies are needed to further clarify the mechanism of action and verify the findings of animal experiments.

In summary, taurine deficiency is closely related to the onset of neurodevelopmental disorders, and dietary supplementation may have a certain therapeutic effect. This study is based on this starting point to propose the basis of project. This study intends to conduct an exploratory randomized, double-blind controlled trial to compare and analyze the effect of taurine supplementation on the improvement of core symptoms in ASD children who were treated with routine behavioral rehabilitation combined with taurine supplement (experimental group) and behavioral rehabilitation combined with placebo (control group) for 3 months and continued follow-up for 12 months. The possible mechanism of action was investigated by detecting intestinal symptoms, intestinal flora, markers of oxidative stress and clinical symptoms of ASD. The aim of this study is to explore an effective and reliable adjuvant therapy for children with ASD. To investigate the curative effect of taurine supplementation on the core symptoms of children with ASD spectrum disorder. To observe the incidence of adverse reactions of taurine supplementation, evaluate the clinical application value of taurine supplementation, and provide theoretical support for further tests.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2.5-18 years at enrollment.
* Meet the diagnosis criteria of ASD by the diagnostic and statistical manual of mental disorders(DSM-5).

Exclusion Criteria:

* Rett behavioral sign, cerebral palsy, other congenital diseases, associated with other inherited metabolic behavioral signs, epilepsy.
* Children who have had an acute or chronic infectious disease in the past 3 months.
* Children with abnormal liver and kidney function, chronic pulmonary heart disease.
* Children who have taken taurine supplements or medications in the past 3 months.
* Parents or patients refuse to participate in the study.
* The investigator determines that the subject is unable to comply with the study requirements.

Ages: 30 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Score of Autism Treatment Evaluation Checklist (ATEC) | From baseline till the 3th month.
  Autism Treatment Evaluation Checklist (ATEC) will be used to evaluate the rehabilitation of ASD core syndromes after interventions, which includes communication, social, perception skills and healthy behaviors. ATEC will be self-assessed by guardians.Severity grading: mild (initial ATEC score 20-49), moderate (initial ATEC score 50-79), severe (initial ATEC score >80). The lower the ATEC scores, the better the rehabilitation.

SECONDARY OUTCOMES:
Score of Autism Treatment Evaluation Checklist (ATEC) | From baseline till the 1st,2rd,6th,9th,12th month.
  Autism Treatment Evaluation Checklist (ATEC) will be used to evaluate the rehabilitation of ASD core syndromes after interventions, which includes communication, social, perception skills and healthy behaviors. ATEC will be self-assessed by guardians.Severity grading: mild (initial ATEC score 20-49), moderate (initial ATEC score 50-79), severe (initial ATEC score >80). The lower the ATEC scores, the better the rehabilitation.
Childhood Autism Rating Scale(CARS) | At the 3rd,6th,9th,12th month from baseline.
  The Childhood Autism Rating Scale (CARS) developed by Schoplen(1980).The total score is 60 points, and CARS will be evaluated by clinicians. Participants with a score15-30,31-36,37-60 are considered as mild autism, moderate autism, severe autism.
6-item Gastrointestinal Severity Index(6-GSI) | At the1st,2rd,3rd,6th,9th,12th month from baseline.
  6-item Gastrointestinal Severity Index(6-GSI) will be used to assess the Gastrointestinal syndromes of ASD patients, including constipation, diarrhea, average stool consistency, stool smell, flatulence, abdominal pain. The higher the score, the more severe the syndromes.
Autism Spectrum Rating Scales(ASRS) | At the1st,2rd,3rd,6th,9th,12th month from baseline.
  The Autism Spectrum Rating Scales (ASRS), consisting of 71 questions, consists of three core parts: defects in the nature of social interaction, abnormalities in language and communication, stereotypes, limitations, and repetitive interests and behaviors.
  ASRS will be self-assessed by guardians. The ASRS questionnaire uses a 5-level score: 0 = never, meaning that it has never happened; 1 point = very few, refers to 1 or 2 times in a month; 2 points = sometimes, refers to 1 or 2 times in a week; 3 points = frequent, meaning 3 or 4 times in a week; 4 points = always, which means every day.
Social Responsiveness Scale(SRS) | At the1st,2rd,3rd,6th,9th,12th month from baseline.
  Social Responsiveness Scale (SRS), which quantifies children's social ability, are used to assess children's social ability. SRS will be self-assessed by guardians. There are five subscales: Social Awareness, Social Cognition, Social Communication and Social motivation And Autistic Mannerisms. The main feature of this scale is to evaluate the social situation of children closely with social disorder as the core symptom of ASD.
Identification and Management of Feeding Difficulties(IMFeD) | At the1st,2rd,3rd,6th,9th,12th month from baseline.
  Identification and Management of Feeding Difficulties(IMFeD), it is composed of 17 items and contains six dimensions: poor appetite, particular food preferences, poor eating habits, excessive parental concern, fear of eating, and underlying disease status. IMFeD will be self-assessed by guardians. The severity of children's eating behavior problems is divided into four levels: "Always" refers to an average of 5 or more days per week when the eating behavior or feeling."Often" means having this behavior or feeling on average 3 to 4 days per week."Sometimes" means having this behavior or feeling on average 1 to 2 days per week."Never" means that the action or feeling does not occur.
Gesell Developmental Scale | At the 3rd,6th,9th,12th month from baseline.
  The Gesell developmental scale mainly assesses the function of the central nervous system. It has five specific domains, gross motor, fine motor, language and individual-social behavior. Gesell Developmental Scale will be evaluated by clinicians.According to the relationship between the scores obtained in 5 behavioral fields and actual age, the development quotient(DQ) of each field was calculated. Edge state: 76≤DQ≤85; Mild stunting: 55≤DQ≤75; Moderate stunting: 40≤DQ≤54; Severe stunting: 25≤DQ≤39; Very severe stunting: DQ<25.
Children's Sleep Habits Questionnaire (CSHQ) | At the1st,2rd,3rd,6th,9th,12th month from baseline.
  Children's Sleep Habits Questionnaire (CSHQ), which contains 48 items, can detect eight specific sleep problems, such as bad sleeping habits, sleep anxiety, irregular sleep duration, sleep disordered breathing, abnormal sleep, daytime sleepiness, night waking, and prolonged sleep latency. CSHQ will be self-assessed by guardians. The CSHQ asked parents to recall their children's sleep conditions in the past four weeks, and rated the children's sleep conditions as "often" (5-7 times per week), "sometimes" (2-4 times per week), and "rarely or none" (0-1 times per week).
The Wechsler intelligence scale (WISC) score | At the 3rd,6th,9th,12th month from baseline.
  WISC consists of 6 verbal subtests, namely general knowledge, similarity, arithmetic, vocabulary, comprehension, and number memorization. WISC will be evaluated by professional clinicians, including 6 operation sub-tests, namely picture complement, picture arrangement, building block pattern, object matching, decoding, maze. A score of ≥130 is very excellent, 120 to 129 is excellent, 110 to 119 is upper middle, 90 to 109 is medium, 80 to 89 is lower middle, 70 to 79 is marginal, < 70 is low intelligence, of which 55 to 69 are mild mental retardation, 40 to 54 are moderate mental retardation, and 25 to 39 are severe mental retardation.

OTHER OUTCOMES:
Change of hemoglobin concentration in cortical metabolism | At the 3rd month from baseline.
  Functional near-infrared spectroscopy (fNIRS) is a new non-invasive neuroimaging technique for real-time monitoring of brain function. Based on the difference of absorption rate of oxygenated hemoglobin (HbO) and deoxyhemoglobin (DHb) in brain tissue for NIR light of different wavelengths, the changes of hemoglobin concentration in cortical metabolism will be calculated to reflect changes of brain function.
Change of taurine-related serum metabolites levels | At the 3rd month from baseline.
  Non-targeted metabolomics analysis will be performed to assess change in several taurine-related serum metabolites levels between group.
Difference in proportions of Intestinal flora species(%) | At the 3rd month from baseline.
  Metagenomics using stool samples will be performed to evaluate intestinal flora diversity between group. The proportion of intestinal flora species(%) will be summarized between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Zhou, Principal Investigator — Guizhou Provincial People's Hospital
Locations (1):
- Guizhou Provincial People's Hospital, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Y, He W, Deng Q, Peng Z, Tai Z, Ma Y, Wang T, Wang Y, Yan W, Zhou H. Taurine supplementation in children with autism spectrum disorders: a study protocol for an exploratory randomized, double-blind, placebo-controlled trial. BMC Pediatr. 2025 Oct 27;25(1):871. doi: 10.1186/s12887-025-06216-0. PMID 41146076

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-02-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT05980520/SAP_000.pdf